CLINICAL TRIAL: NCT01053741
Title: The Effect of Seminal Fluid on Distal Colon Mucosal Permeability and Susceptibility to HIV Infection
Brief Title: Effect of Seminal Fluid on the Colon Wall; Implications for HIV Transmission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NA_00014051
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seminal Fluid then Normosol (Experimental): 2.5 mL radiolabeled autologous seminal fluid administered rectally x1. Two week pause between interventions. Then 2.5 mL radiolabeled Normosol-R administered rectally X1.
  Interventions: Biological: Radiolabeled autologous seminal fluid; Biological: Radiolabeled Normosol-R
- Normosol then Seminal Fluid (Experimental): 2.5 mL radiolabeled Normosol-R administered rectally x1. Two week pause between interventions. Then 2.5 mL radiolabeled autologous seminal fluid administered rectally X1.
  Interventions: Biological: Radiolabeled autologous seminal fluid; Biological: Radiolabeled Normosol-R

INTERVENTIONS:
Biological: Radiolabeled autologous seminal fluid — Autologous lymphocytes labeled with 250 microcuries In-111 and 500 microcuries Tc-99m in seminal fluid vehicle.
Biological: Radiolabeled Normosol-R — Autologous lymphocytes labeled with 250 microcuries In-111 and 500 microcuries Tc-99m in Normosol-R fluid vehicle.

SUMMARY:
This research is being done to learn how seminal fluid affects the lining of the colon, and whether this might make it easier for HIV to get into the body and cause infection.

DETAILED DESCRIPTION:
Design of effective rectal microbicides to prevent HIV infection requires an understanding of rectal HIV transmission and the location within the lower gastrointestinal (GI) tract (luminal and mucosal) of HIV (cell-free and cell-associated) following exposure to infected seminal fluid. These basic details of HIV transmission have yet to be determined in human subjects, yet they are essential to select microbicide candidates if they are to be rationally designed to achieve effective concentrations at sites of HIV transmission. Rational development of a rectal microbicide also requires an understanding of those factors that may contribute to colonic mucosal injury - potential confounders of microbicidal effect. Such factors include exposure to seminal fluid which has been shown in animal and in vitro studies to cause histologic and permeability changes that might facilitate HIV transmission.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed informed consent
* Men of 21 years or older.
* Prior history of receptive anal intercourse.
* Laboratory values within the last 28 days:
* Negative for HIV antibodies
* Lymphocyte count within normal limits
* Neutrophil count > 1,000 cells/ml
* Cluster of Differentiation 4 (CD4) cell count > 500 cells/ml
* Platelet count ≥ 150,000 cells/mm3
* Prothrombin Time (PT) within normal limits
* Partial thromboplastin time (PTT) within normal limits.
* No childbearing intentions.

Exclusion Criteria:

* Active anorectal disease or recent (3 months) anorectal surgery;
* Diarrhea, defined as three or more loose stools per day, for at least three days prior to admission.
* History of sleep apnea, or airway problems with previous sedation procedures.
* History of significant adverse reaction to sedation medications.
* Other history, including significant occupational radiation exposure, history of inflammatory bowel disease or any other diseases and lab results, such that, in the judgment of the investigator, study procedures are not considered safe for the subject's participation.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Fuchs, PA-C, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Drug Development Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is an exploratory physiologic study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment initiated September 2008, completed October 2009. Study participants recruited from previous trial participation and advertisements posted in the medical institutions.
Groups:
- Seminal Fluid, Then Normosol-R: Subjects first received 2.5 mL radiolabeled autologous seminal fluid administered rectally x1. Than a two week pause between interventions. Followed by 2.5 mL radiolabeled Normosol-R administered rectally x1.
- Normosol-R Then Seminal Fluid: Subjects first received 2.5 mL radiolabeled Normosol-R administered rectally x1. Then a two week pause between interventions. Followed by 2.5 mL radiolabeled autologous seminal fluid administered rectally x1.
Period: 1st Intervention
Arm/Group | Seminal Fluid, Then Normosol-R | Normosol-R Then Seminal Fluid
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: 14 Day Washout
Arm/Group | Seminal Fluid, Then Normosol-R | Normosol-R Then Seminal Fluid
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: 2nd Study Intervention
Arm/Group | Seminal Fluid, Then Normosol-R | Normosol-R Then Seminal Fluid
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Normosol-R Then Seminal Fluid: 2.5 mL radiolabeled Normosol-R administered rectally x1. Two week pause between interventions. Then 2.5 mL radiolabeled autologous seminal fluid administered rectally X1.
  Radiolabeled autologous seminal fluid: Autologous lymphocytes labeled with 250 microcuries In-111 and 500 microcuries Tc-99m in seminal fluid vehicle.
  Radiolabeled Normosol-R: Autologous lymphocytes labeled with 250 microcuries In-111 and 500 microcuries Tc-99m in Normosol-R fluid vehicle.
- Total: Total of all reporting groups
Arm/Group | Seminal Fluid Then Normosol | Normosol-R Then Seminal Fluid | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Full Range); unit: years] | 44 [34 to 50] | 40 [21 to 48] | 41.5 [21 to 50]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male gender | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Epithelial Disruption Graded by a Pathologist Blinded to Study Intervention.
Description: Endoscopy will be performed to obtain biopsy specimens at baseline and following each inpatient enema exposure. Samples will be obtained at each flexible sigmoidoscopy and set aside for batch sectioning and H&E staining. Slides will be reviewed and scored by a qualified pathologist blinded to treatment assignment using a qualitative scoring system. This scoring system uses semi-quantitative scoring that focuses on acute toxicity to epithelial cell layer similar to that seen in animal studies. This is a categorical grading scale, where 0 = Epithelial surface intact;1 = <1/3 of surface denuded; 2 = 1/3 - 2/3rds of surface denuded;3 = More than 2/3rds of surface denuded.
  Six separate biopsies for each subject and each treatment intervention were analyzed in a multi-level analysis. In comparison with the baseline condition (no intervention), the odds and 95% confidence interval (CI) of having a higher epithelial denudation score were calculated for each intervention.
Time Frame: One hour
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Seminal Fluid: Seminal Fluid Intervention
- Normosol-R: Normosol-R Intervention
Arm/Group | Seminal Fluid | Normosol-R
Number analyzed (Participants) | 10 | 10
units on a scale | 1.0 [0.92 to 1.17] | 1.17 [1.04 to 1.46]
Statistical Analysis 1: Comparison: Seminal Fluid vs Normosol-R; Null hypothesis is that there is no difference in epithelial surface disruption when comparing the two interventions. Power calculation was based on identifying a median difference in histology grade of 0.83, using a two-sided alpha of 0.05 with 90% power in 10 subjects; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Seminal Fluid | Normosol-R
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seminal Fluid (N=10) | Normosol-R (N=10)
Gas/bloating (Gastrointestinal disorders) | 4 (4) | 3 (3) — symptoms following flexible sigmoidoscopy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No